CLINICAL TRIAL: NCT02393586
Title: Evaluating Pharmacokinetics and Whole Blood Bactericidal Activity Against Mycobacterium Tuberculosis of Single Doses of Faropenem Plus Amoxicillin/Clavulanic Acid in Healthy Volunteers
Brief Title: Whole Blood Bactericidal Activity (WBA) Against Mycobacterium Tuberculosis of Faropenem Plus Amoxicillin/Clavulanic Acid in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Faro-WBA
Record Dates: First submitted 2015-03-06; First posted 2015-03-19 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; Whole blood Bactericidal Activity; WBA; Faropenem
MeSH Terms: conditions — Tuberculosis | interventions — fropenem; Amoxicillin; Clavulanic Acid; Amoxicillin-Potassium Clavulanate Combination; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Faropenem/augmentin (Experimental): Faropenem 600mg plus amoxicillin/clavulanic acid 500mg/125mg
  Interventions: Drug: Faropenem; Drug: Amoxicillin/clavulanic acid 500mg/125mg
- Rifampicin/faropenem/augmentin (Experimental): Rifampicin 10mg/kg plus faropenem 600mg plus amoxicillin/clavulanic acid 500mg/125mg
  Interventions: Drug: Faropenem; Drug: Amoxicillin/clavulanic acid 500mg/125mg; Drug: Rifampicin
- Rifampicin (Experimental): Rifampicin 10mg/kg
  Interventions: Drug: Rifampicin

INTERVENTIONS:
Drug: Faropenem — Single oral dose
  Other Names: Faropenem sodium
  Arms: Faropenem/augmentin; Rifampicin/faropenem/augmentin
Drug: Amoxicillin/clavulanic acid 500mg/125mg — Single oral dose
  Other Names: Augmentin
  Arms: Faropenem/augmentin; Rifampicin/faropenem/augmentin
Drug: Rifampicin — Single oral dose
  Other Names: Rifampin
  Arms: Rifampicin; Rifampicin/faropenem/augmentin

SUMMARY:
The purpose of this study is to evaluate the bactericidal activity against Mycobacterium tuberculosis of faropenem boosted with amoxicillin/clavulanic acid. Pharmacokinetics (PK) and Whole blood Bactericidal Activity (WBA) will be measured in healthy volunteers following single doses of faropenem plus amoxicillin/clavulanic acid.

DETAILED DESCRIPTION:
WBA is an ex vivo model for measuring the combined effects of administered drugs, host factors and strain factors on mycobacterial killing. If performed in parallel with PK measurements, the method can be used to evaluate the effect of drugs throughout the dosing cycle. The aim of this trial is to investigate the bactericidal activity of faropenem administered with amoxicillin/clavulanic acid (augmentin) using the WBA model. We will also explore whether there is any additive effect or synergy with rifampicin in this model. The activity of faropenem on WBA by different strains of M. tuberculosis will be compared and the relationship between the host immune profile and WBA will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 21 and above
2. Male or female willing to comply with the study visits and procedures
3. Willing and able to provide written informed consent

Exclusion Criteria:

1. Women who are currently pregnant or breastfeeding
2. Signs of active TB
3. Previous hypersensitivity or allergy to rifampicin, faropenem or other beta-lactam drugs (penicillins, carbapenems)
4. Current use of any drugs or medications known to have an interaction with any of the study drugs
5. Current use of any other drugs, over the counter or herbal preparations that are known or potential inhibitors or inducers of cytochrome P450 enzymes
6. Evidence of renal or hepatic dysfunction or any clinically significant deviation from normal during screening including laboratory determinations
7. Known hepatic disease or alcohol abuse
8. Any other significant condition that would, in the opinion of the investigator, compromise the volunteer's safety or outcome in the trial
9. Current participation in other clinical intervention trial or research protocol

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2015-02; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Cumulative WBA | 8 hours
  Cumulative bactericidal activity (WBA) reported as change in Mtb log CFU per day based on values observed (AUC)

SECONDARY OUTCOMES:
The pharmacokinetic profile of study drug(s) | 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Paton, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Derived] Gurumurthy M, Verma R, Naftalin CM, Hee KH, Lu Q, Tan KH, Issac S, Lin W, Tan A, Seng KY, Lee LS, Paton NI. Activity of faropenem with and without rifampicin against Mycobacterium tuberculosis: evaluation in a whole-blood bactericidal activity trial. J Antimicrob Chemother. 2017 Jul 1;72(7):2012-2019. doi: 10.1093/jac/dkx081. PMID 28333342
- Available data/document: Link to Pubmed (Final publication) — https://www.ncbi.nlm.nih.gov/pubmed/28333342